CLINICAL TRIAL: NCT03896724
Title: A Phase Ib/IIb Randomised Controlled Trial of the Safety, Immunogenicity and Efficacy of a Candidate Malaria Vaccine, R21 Adjuvanted With Matrix-M (R21/MM), in 5-17 Month Old Children in Nanoro, Burkina Faso
Brief Title: Safety, Immunogenicity and Efficacy of R21 Matrix-M in 5-17 Month Old Children in Nanoro, Burkina Faso
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAC076
Record Dates: First submitted 2019-01-18; First posted 2019-04-01 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Matrix-M; Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): n=150. Age 5-17 month-old. 5mcg R21/25mcg Matrix-M at Day 0, 28 and 56 and 1 year.
  Following the initial booster, Group 1 will be randomised 2:1 into Groups1a and 1b for 5ug R21/50ug Matrix-M: control. Groups 1a and 1b will receive these second and third booster vaccinations each year prior to the malaria season
  Interventions: Biological: R21 adjuvanted with 25mcg Matrix-M; Biological: Rabies Vaccine; Biological: R21 adjuvanted with 50mcg Matrix-M
- Group 2 (Experimental): n=150. Age 5-17 month-old. 5mcg R21/50mcg Matrix-M at Day 0, 28 and 56 and 1 year.
  Following the initial booster, Group 2 will be randomised 2:1 into Groups 2a and 2b or 5ug R21/50ug Matrix-M:ccontrol. Groups 2a and 2b will receive these second and third booster vaccinations each year prior to the malaria season
  Interventions: Biological: Rabies Vaccine; Biological: R21 adjuvanted with 50mcg Matrix-M
- Group 3 (control group) (Placebo Comparator): n=150. Age 5-17 month-old. Rabies Vaccine by the end of the trial.
  Interventions: Biological: Rabies Vaccine

INTERVENTIONS:
Biological: R21 adjuvanted with 25mcg Matrix-M — Vaccine
  Arms: Group 1
Biological: Rabies Vaccine — Vaccine
Biological: R21 adjuvanted with 50mcg Matrix-M — vaccine
  Arms: Group 1; Group 2

SUMMARY:
This is a double blind randomised controlled clinical trial to evaluate the efficacy of R21 adjuvanted with Matrix-M in healthy 5-17 month old children in a malaria endemic area.

DETAILED DESCRIPTION:
In this double-blind, randomised, controlled, phase 2b trial, the low-dose circumsporozoite protein-based vaccine R21, with two different doses of adjuvant Matrix-M (MM), was given to children aged 5-17 months in Nanoro, Burkina Faso-a highly seasonal malaria transmission setting. Three vaccinations were administered at 4-week intervals before the malaria season, with a fourth dose 1 year later. All vaccines were administered intramuscularly into the thigh. Group 1 received 5 μg R21 plus 25 μg MM, group 2 received 5 μg R21 plus 50 μg MM, and group 3, the control group, received rabies vaccinations. Children were randomly assigned (1:1:1) to groups 1-3. An independent statistician generated a random allocation list, using block randomisation with variable block sizes, which was used to assign participants. Participants, their families, and the local study team were all masked to group allocation. Only the pharmacists preparing the vaccine were unmasked to group allocation. Vaccine safety, immunogenicity, and efficacy were evaluated over 1 year. The primary objective assessed protective efficacy of R21 plus MM (R21/MM) from 14 days after the third vaccination to 6 months.

From May 7 to June 13, 2019, 498 children aged 5-17 months were screened, and 48 were excluded. 450 children were enrolled and received at least one vaccination. 150 children were allocated to group 1, 150 children were allocated to group 2, and 150 children were allocated to group 3. The final vaccination of the primary series was administered on Aug 7, 2019. R21/MM had a favourable safety profile and was well tolerated.

Please see publication for more details: Lancet. 2021 May 15;397(10287):1809-1818. doi: 10.1016/S0140-6736(21)00943-0

After the first booster vaccination, participants in Groups 1 and 2 were further randomised 2:1 to receive R21 with Matrix-M: control. The trial was extended by a further two years with yearly boosters of R21/MM or rabies vaccine. Groups 1 and 2 were subdivided and randomized 2:1 to receive R21/MM or rabies vaccine as the second booster. Group 3 received control rabies vaccine as they had done previously. The second boosting occurred between June and July 2021 where 368 participants were boosted. In May 2022 it was decided to amend the protocol to allow for groups 1a and 2a (malaria vaccine groups) to be randomised 1:1 to receive either the R21/Matrix-M vaccine or a control rabies vaccine a year after the previous booster vaccine. The third boosting occurred between June and July 2022 where 357 participants were boosted.

Between June 2, and July 2, 2020, 409 children returned to receive a booster vaccine. Each child received the same vaccination for the booster as they received in the primary series of vaccinations; 132 participants received 5 μg R21 adjuvanted with 25 μg Matrix-M, 137 received 5 μg R21 adjuvanted with 50 μg Matrix-M, and 140 received the control vaccine.

A booster dose of R21/Matrix-M at 1 year following the primary three-dose regimen was administered. The trial is ongoing to assess long-term follow-up of these participants and the value of further booster

Please see publication for more details of results of two year follow up: Lancet Infect Dis. 2022 Dec;22(12):1728-1736. doi: 10.1016/S1473-3099(22)00442-X.

VAC076 is complete, with the last volunteer last visit occurring in July 2023. This trial was funded by the European and Developing Countries Clinical Trials Partnership (reference: RIA2016V-1649 MMVC).

ELIGIBILITY:
Inclusion Criteria:

* Healthy child aged 5-17 months at the time of first study vaccination
* Provide written Informed consent of parent/guardian
* Child and parent/guardian resident in the study area villages and anticipated to be available for vaccination and follow-up for 2 years following last dose of vaccination

Exclusion Criteria:

* Clinically significant skin disorder (psoriasis, contact dermatitis etc.), immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness.
* Weight-for-age Z score of less than -3 or other clinical signs of malnutrition.
* History of allergic reaction, significant IgE-mediated event, or anaphylaxis to immunisation.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, e.g. neomycin.
* Sickle cell disease.
* Clinically significant laboratory abnormality as judged by the study clinician.
* Blood transfusion within one month of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Previous vaccination with experimental malaria vaccines.
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Current participation in another clinical trial, or within 12 weeks of this study.
* Known maternal HIV infection (No testing will be done by the study team).
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (For corticosteroids, this will mean prednisone, or equivalent, >= 0.5 mg/kg/day. Inhaled and topical steroids are allowed).
* Any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 5 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
The protective efficacy (number of cases) against clinical malaria of R21 adjuvanted with Matrix-M in 5-17 month old children living in a malaria-endemic area | for 6 months after the last vaccination
  We will look for the presence of axillary temperature ≥37.5°C AND P. falciparum parasites density > 5000 asexual forms/µL as a primary case definition of clinical malaria.
  - We will look for the presence of axillary temperature ≥37.5°C and/ or history of fever within the last 24 hours AND P. falciparum parasites density > 0 for a secondary case definition of clinical malaria.

SECONDARY OUTCOMES:
Duration of Protective efficacy (number of cases) against clinical malaria | for 12 months after administration of the third dose of vaccine, and for 6 and 12 months after each booster vaccination
  To assess the protective efficacy (number of cases) against clinical malaria of R21 adjuvanted with Matrix-M in 5-17 months old children living in a malaria-endemic area
Efficacy (number of cases) against asymptomatic P. falciparum infection | at 6 and 12 months after administration of the third dose of vaccine, and for 12 months after each booster vaccination
  Primary case definition of asymptomatic P. falciparum infection: Presence of axillary temperature < 37.5°C and absence of history of fever within the last 24 hours; AND P. falciparum parasites density > 0 asexual forms/µL
The safety and reactogenicity (number of adverse events) of R21 adjuvanted with Matrix-M in 5-17 month olds living in a malaria-endemic area in the month following each vaccination and at 12 months after administration of the final dose of vaccine | for 6 and 12 months after administration of the third dose of vaccine, and for 12 months after each booster vaccination
  * Occurrence of solicited local and/or systemic reactogenicity signs and symptoms for 7 days following the vaccination
  * Occurrence of unsolicited adverse events for 28 days following the vaccination
  * Occurrence of serious adverse events for the duration of the trial
The humoral immunogenicity (antibody response) of R21 adjuvanted with Matrix-M in 5-17 months old children living in a malaria-endemic area | for 6 and 12 months after administration of the third dose of vaccine, and for 6 months after each booster vaccination
  * Comparison of immunogenicity (antibody responses to CSP) in the R21/MM vaccination group with those in the rabies vaccine group and the durability of responses
  * ELISA to quantify antibodies to the vaccine components (regions of the CS antigen including the NANP repeat region and other elements of the protein as well as anti HBs).

OTHER OUTCOMES:
Exploratory Objectives: Efficacy (number of cases) against incident cases of severe malaria | 12 months after administration of the final dose of vaccine
  Primary case definition of severe malaria:
  Presence of P. falciparum parasites density > 5000 asexuals forms/µL; AND one of more of the following criteria of disease severity:
  * Prostration
  * Respiratory distress
  * Blantyre coma score ≤ 3
  * Seizures: 2 or more
  * Hypoglycemia < 2.2 mmol/L
  * Acidosis BE ≤-8.0 mmol/L
  * Lactate ≥ 5.0 mmol/L
  * Anemia < 5.0 g/dL
  * Acute kidney injury
  * Pulmonary oedema
  * Significant bleeding
  * Shock (systolic BP <70mm Hg); AND
    -Without any of the following criteria of co- morbidity
  * Pneumonia (confirmed by X-ray)
  * Meningitis (confirmed by CSF examination)
  * Sepsis (with Positive blood culture)
  * Gastroenteritis with dehydration
Exploratory Objectives: Gut microbiome (bacterial communities identified) effect on vaccine response. | for 12 months after administration of the final dose of vaccine
  • DNA extraction and sequencing to determine differences in gut microbiome between those who respond to vaccination and those who don't.
Exploratory Objectives: Genetic testing to elicit differences in vaccine response. | for 12 months after administration of the final dose of vaccine
  * Genetic tests-determination of human HLA-type and genotyping of any other genes to assess impact on response to vaccination, including genome-wide SNP and sequence analysis.
  * Genetic testing of the DNA of malaria parasites identified during the study to determine if the vaccine preferentially protects against specific genetic types of P. falciparum.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche en Sciences de la Sante - Clinical Research Unit of Nanoro (IRSS-URCN), Nanoro, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Study information will be made available through an open repository. The information to be made available will be anonymized so that there is no link to participants and will include data on safety, immune responses and any other data generated from samples obtained in this study.
Supporting Information: Study Protocol, SAP
Time Frame: Within 12 months of manuscripts related to the trial being published.
Access Criteria: A link to the data respository will be given below

REFERENCES:
- [Derived] Mukhopadhyay ES, Bellamy DG, Tinto H, Hamaluba M, Truby A, Salman AM, Hill AVS. Naturally acquired immune responses to alpha-gal in malaria endemic settings and pre-clinical efficacy testing with R21/MM. Vaccine. 2025 Dec 5;68:127897. doi: 10.1016/j.vaccine.2025.127897. Epub 2025 Nov 1. PMID 41176969
- [Derived] Datoo MS, Natama HM, Some A, Bellamy D, Traore O, Rouamba T, Tahita MC, Ido NFA, Yameogo P, Valia D, Millogo A, Ouedraogo F, Soma R, Sawadogo S, Sorgho F, Derra K, Rouamba E, Ramos-Lopez F, Cairns M, Provstgaard-Morys S, Aboagye J, Lawrie A, Roberts R, Valea I, Sorgho H, Williams N, Glenn G, Fries L, Reimer J, Ewer KJ, Shaligram U, Hill AVS, Tinto H. Efficacy and immunogenicity of R21/Matrix-M vaccine against clinical malaria after 2 years' follow-up in children in Burkina Faso: a phase 1/2b randomised controlled trial. Lancet Infect Dis. 2022 Dec;22(12):1728-1736. doi: 10.1016/S1473-3099(22)00442-X. Epub 2022 Sep 7. PMID 36087586
- [Derived] Datoo MS, Natama MH, Some A, Traore O, Rouamba T, Bellamy D, Yameogo P, Valia D, Tegneri M, Ouedraogo F, Soma R, Sawadogo S, Sorgho F, Derra K, Rouamba E, Orindi B, Ramos Lopez F, Flaxman A, Cappuccini F, Kailath R, Elias S, Mukhopadhyay E, Noe A, Cairns M, Lawrie A, Roberts R, Valea I, Sorgho H, Williams N, Glenn G, Fries L, Reimer J, Ewer KJ, Shaligram U, Hill AVS, Tinto H. Efficacy of a low-dose candidate malaria vaccine, R21 in adjuvant Matrix-M, with seasonal administration to children in Burkina Faso: a randomised controlled trial. Lancet. 2021 May 15;397(10287):1809-1818. doi: 10.1016/S0140-6736(21)00943-0. Epub 2021 May 5. PMID 33964223